CLINICAL TRIAL: NCT03769467
Title: An Open-Label Phase 1B/2 Study to Evaluate the Safety and Efficacy of Tabelecleucel in Combination With Pembrolizumab in Subjects With Platinum-pretreated, Recurrent/Metastatic Epstein-Barr Virus-Associated Nasopharyngeal Carcinoma
Brief Title: Tabelecleucel in Combination With Pembrolizumab in Subjects With Epstein-Barr Virus-associated Nasopharyngeal Carcinoma (EBV+ NPC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Phase 1B part was completed with review of DLTs and cumulative safety data by Safety Data Review Committee and identification of a safe RP2D. Post-internal review, sponsor decided to terminate the study, and hence, Phase 2 part was not conducted.
Sponsor: Atara Biotherapeutics (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATA129-NPC-202; KEYNOTE PN597 (Other: Merck Sharp & Dohme Corp.)
Record Dates: First submitted 2018-11-29; First posted 2018-12-07 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-09

CONDITIONS: Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms; Epstein-Barr Virus Infections; Epstein-Barr Viraemia; Epstein-Barr Virus-associated Nasopharyngeal Carcinoma (EBV+ NPC)
Keywords: Nasopharyngeal Carcinoma (NPC); NPC; Nasopharyngeal Cancer; Nose Cancer; Epstein-Barr Virus (EBV); Epstein-Barr Virus Viremia; EBV-associated NPC; Allogeneic, off-the-shelf T-cell; immunotherapy; Head and Neck Cancer; Carcinoma; Nasopharyngeal Neoplasms; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Pharyngeal Neoplasms; Otorhinolaryngologic Neoplasms; Head and Neck Neoplasms; Neoplasms by Site; Nasopharyngeal Diseases; Pharyngeal Diseases; Stomatognathic Diseases; Otorhinolaryngologic Diseases; Pembrolizumab; Programmed death-1 (PD-1); Programmed death-ligand 1(PD-L1)
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Nasopharyngeal Neoplasms; Epstein-Barr Virus Infections; Nose Neoplasms; Head and Neck Neoplasms; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Pharyngeal Neoplasms; Otorhinolaryngologic Neoplasms; Neoplasms by Site; Nasopharyngeal Diseases; Pharyngeal Diseases; Stomatognathic Diseases; Otorhinolaryngologic Diseases | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1B: Checkpoint Inhibitor Naïve (Experimental): Checkpoint inhibitor naive subjects during the treatment phase will receive intravenous (IV) infusion of pembrolizumab at 200 mg for adults (≥ 18 years of age) or 2 mg/kg for adolescents (12 to < 18 years of age) prior to the administration of tabelecleucel on Day 1; and IV infusion of tabelecleucel (tab-cel) at 2 × 10^6 T-cells/kg on Days 1, 8, and 15 of each 21-day treatment/consolidation cycles (at least 2 cycles or up to 4 cycles). From the Maintenance Phase, subjects with stable disease or better will receive tabelecleucel on Day 1 and pembrolizumab on Day 1, Day 21, Day 42, and Day 63 of each 84- day maintenance cycle, which was continued until disease progression, unacceptable toxicity, or a total of 35 pembrolizumab infusions (including for treatment, consolidation, and maintenance) had been administered, whichever occurred first.
  Interventions: Biological: Tabelecleucel; Biological: Pembrolizumab
- Cohort 1B: Checkpoint Inhibitor PD-1/PD-L1 Failure (Experimental): Checkpoint inhibitor PD-1/PD-L1 failure subjects during the treatment phase will receive IV infusion of pembrolizumab at 200 mg for adults (≥ 18 years of age) or 2 mg/kg for adolescents (12 to < 18 years of age) prior to the administration of tabelecleucel on Day 1; and IV infusion of tabelecleucel (tab-cel) at 2 × 10^6 T-cells/kg on Days 1, 8, and 15 of each 21-day treatment/consolidation cycles (at least 2 cycles or up to 4 cycles).). From the Maintenance Phase, subjects with stable disease or better will receive tabelecleucel on Day 1 and pembrolizumab on Day 1, Day 21, Day 42, and Day 63 of each 84-day maintenance cycle, which was continued until disease progression, unacceptable toxicity, or a total of 35 pembrolizumab infusions (including for treatment, consolidation, and maintenance) had been administered, whichever occurred first.
  Interventions: Biological: Tabelecleucel; Biological: Pembrolizumab
- Cohort 2: Checkpoint Inhibitor Naïve (Experimental): Checkpoint inhibitor naive subjects during the treatment phase will receive IV infusion of pembrolizumab at 200 mg for adults (≥ 18 years of age) or 2 mg/kg for adolescents (12 to < 18 years of age) prior to the administration of tabelecleucel on Day 1; and IV infusion of tabelecleucel (tab-cel) at 2 × 10^6 T-cells/kg on Days 1, 8, and 15 of each 21-day treatment/consolidation cycles (at least 2 cycles or up to 4 cycles). From the Maintenance Phase, subjects with stable disease or better will receive tabelecleucel on Day 1 and pembrolizumab on Day 1, Day 21, Day 42, and Day 63 of each 84- day maintenance cycle, which was continued until disease progression, unacceptable toxicity, or a total of 35 pembrolizumab infusions (including for treatment, consolidation, and maintenance) had been administered, whichever occurred first.
  Interventions: Biological: Tabelecleucel; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Tabelecleucel — Tabelecleucel is an off-the-shelf, allogeneic T-cell immunotherapy for the treatment of EBV+ malignancies and diseases.
  Other Names: tab-cel®; ATA129; Epstein-Barr Virus-specific Cytotoxic T Lymphocytes (EBV-CTL)
Biological: Pembrolizumab — pembrolizumab IV infusion
  Other Names: MK-3475

SUMMARY:
This is a multicenter, open-label, single-arm Phase 1B/2 study to assess the safety and efficacy of tabelecleucel in combination with pembrolizumab for the treatment of subjects with platinum-pretreated, recurrent/metastatic Epstein-Barr Virus-associated Nasopharyngeal Carcinoma (EBV+ NPC).

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm Phase 1B/2 study to assess the safety and efficacy of tabelecleucel in combination with pembrolizumab for the treatment of subjects with platinum-pretreated, recurrent/metastatic EBV+ NPC.

Tabelecleucel will be selected for each subject from the bank of available tabelecleucel cell products based on matching ≥ 2 human leukocyte antigen (HLA) alleles, at least one of which is a restricting HLA allele, shared between the tabelecleucel donor and the subject's EBV+ NPC. Sites will provide high resolution HLA typing of the subject and other information as required by the protocol.

Phase 1B will identify the maximum tolerated dose (MTD) and characterize the dose limiting toxicity (DLT) for tabelecleucel in combination with pembrolizumab in up to 24 subjects. In the absence of an MTD, the recommended Phase 2 dose (RP2D) will be identified. Phase 2 will evaluate the safety and efficacy of the combination in 36 subjects at the recommended dose level from Phase 1B.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 12 years of age.
2. Incurable, locally recurrent or metastatic Epstein-Barr virus (EBV)+NPC (World Health Organization type II/III) in whom the EBV nucleic acid or antigens have been demonstrated in tissue biopsy samples.
3. Subjects must have had prior receipt of platinum-containing regimen either:

   1. For the treatment of recurrent or metastatic disease, or
   2. Experienced progression of disease within 6 months following completion of a platinum-based combination therapy as part of (neo)adjuvant chemotherapy. Note: Subject who had only concurrent chemoradiation therapy without (neo)adjuvant therapy and then recurred/metastasized must have progressed on at least 1 platinum-containing regimen for their recurrent/metastatic disease before study entry.
4. Phase 1B (Cohort 1):

   1. Checkpoint inhibitor naïve (have never received pembrolizumab or any other anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-OX40 or anti-CTLA-4 antibodies) OR
   2. Refractory to an anti-programmed cell death protein-1 (PD-1) or anti-programmed death-ligand1 (PD-L1) monoclonal antibody approved by the local regulatory agency either as monotherapy or in combination with other checkpoint inhibitors or therapies according to their approved label. To be considered refractory to an anti-PD-1 or anti-PD-L1 monoclonal antibody, all of the following criteria must be met:

   i. Received at least 2 doses of anti-PD-1 or anti-PD-L1 monoclonal antibody at a local regulatory agency-approved dose and schedule. ii. Have progressive disease after anti-PD-1 or anti-PD-L1 monoclonal antibody as defined according to Response Evaluation Criteria in Solid Tumors) RECIST 1.1. The initial evidence of progressive disease is to be confirmed by a second assessment, no less than 4 weeks from the date of the first documented progressive disease, in the absence of rapid clinical progression. (The eligibility determination will be made by the investigator and then the sponsor will collect for retrospective analysis at a central vendor. Once progressive disease is confirmed, the initial date of progressive disease documentation will be considered the date of disease progression).

   iii. Documented disease progression within 24 weeks of the last dose of anti-PD-1 or anti-PD-L1 monoclonal antibody. A subject who was re-treated with anti-PD-1 or anti-PD-L1 monoclonal antibody and a subject who was on maintenance with an anti-PD-1 or anti-PD-L1 monoclonal antibody will be allowed to enter the study as long as there is documented PD within 24 weeks of the last treatment date (with the anti-PD-1 or anti-PD-L1 monoclonal antibody).
5. Phase 1B (Cohort 1): If PD-1/PD-L1 failure (ie, refractory to or relapsed after PD-1/PD-L1 treatment), must have a lesion that can be biopsied after administration of tabelecleucel with acceptable clinical risk (as judged by the investigator) and must agree to undergo biopsy before Cycle 1 Day 1.
6. Phase 2 (Cohort 2): Checkpoint inhibitor naïve (have never received pembrolizumab or any other anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-OX40 or anti-CTLA-4 antibodies).
7. For all subjects: Agree to submit prior biopsy material, if available, for biomarker assessment.
8. Life expectancy ≥ 4 months at time of screening.
9. Measurable disease using RECIST 1.1. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been documented in such lesions.
10. Eastern Cooperative Oncology Group (ECOG) performance status of < 2 for subjects aged > 16 years; Lansky score ≥ 70 for subjects aged 12 to 16 years.
11. Adequate organ function per the protocol.
12. Willing and able to provide written informed consent (pediatric subjects 12 to < 18 years of age must provide assent along with consent from the subject's legally authorized representative).

Exclusion Criteria:

1. Disease that is suitable for local therapy administered with curative intent.
2. Requires vasopressor or ventilator support.
3. Received antithymocyte globulin or similar anti-T-cell antibody therapy ≤ 4 weeks prior to Cycle 1 Day 1.
4. Diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to Cycle 1 Day 1 of study treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the sponsor's medical monitor.
5. Active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
6. History or evidence of interstitial lung disease.
7. History of severe hypersensitivity (Grade ≥ 3) to pembrolizumab and/or any of its excipients.
8. Active infection requiring systemic therapy.
9. History of (non-infectious) pneumonitis that required steroids or current pneumonitis.
10. Received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including granulocyte-colony stimulating factor, granulocyte macrophage-colony stimulating factor or recombinant erythropoetin) within 4 weeks prior to study Day 1.
11. Unresolved immunotherapy-related AEs or treatment for these events within 4 weeks prior to enrollment.
12. History of severe immunotherapy-related adverse effects (Common Terminology Criteria for Adverse Events [CTCAE] grade 4 or CTCAE grade 3 requiring treatment > 4 weeks).
13. Received any non-oncology vaccine therapy used for prevention of infectious diseases for up to 30 days prior to enrollment. Examples include, but are not limited to: measures, mumps, rubella, chicken pox, yellow fever, rabies, bacille Calmette-Guerin, and typhoid vaccine. Seasonal flu vaccines that do not contain live virus are acceptable.
14. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
15. Pregnancy or breastfeeding: females of childbearing potential must have a negative serum pregnancy test. The serum pregnancy must be confirmed negative within 72 hours of Cycle 1 Day 1 (first dose of investigational product) for the subject to be eligible.
16. Female of childbearing potential or male with a female partner of childbearing potential unwilling to use a highly effective method of contraception (abstinence is acceptable) for the course of the study through 120 days after the last study dose.
17. Inability to comply with study procedures.
18. Received chemotherapy or targeted small molecule therapy within 2 weeks of Cycle 1 Day 1. Subjects must have recovered (ie, grade ≤ 1 or at baseline) from adverse events (AEs) due to a previously administered agent. Subjects with grade ≤ 2 neuropathy or grade ≤ 2 alopecia are an exception to this criterion.
19. Received prior radiotherapy within 2 weeks of Cycle 1 Day 1. Subjects must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1- week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-central nervous system (CNS) disease.
20. Antibody/biologic therapy within 4 weeks of Cycle 1 Day 1 or not recovered (i.e., grade ≤ 1 or at baseline) from AEs due to agents administered more than 4 weeks earlier.
21. Carcinomatous meningitis; and/or active CNS metastases, unless metastases are treated and stable and the subject does not require systemic steroids. NOTE: Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging [using the identical imaging modality for each assessment, either magnetic resonance imaging (MRI) or computed tomography (CT) scan] for at least four weeks prior to the first dose of investigational product and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to first dose of investigational product. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
22. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
23. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
24. Known history of human immunodeficiency virus (HIV), known active hepatitis B virus (HBV; e.g., hepatitis B surface antigen [HBsAg] reactive), or hepatitis C virus (HCV; e.g., HCV ribonucleic acid [RNA] is detected).
25. Prior treatment with any investigational product within 4 weeks of Cycle 1 Day 1.
26. Prior treatment with EBV T cells.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2021-08-19 (Actual); Study Completion 2021-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aditi Mehta, DO, Study Director — Atara Biotherapeutics
Locations (7):
- United States (7):
  - City of Hope, Duarte, California
  - Stanford Hospital and Clinics, Palo Alto, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Atlantic Health System / Morristown Medical Center, Morristown, New Jersey
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania (Adults and Pediatrics), Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 12 participants were enrolled in phase 1b (cohort 1). No participants were enrolled in phase 2 (cohort 2) due to early study termination.
Groups:
- Cohort 1B: Checkpoint Inhibitor Naïve: Checkpoint inhibitor naive subjects during the treatment phase received intravenous (IV) infusion of pembrolizumab at 200 mg for adults (≥ 18 years of age) or 2 mg/kg for adolescents (12 to < 18 years of age) prior to the administration of tabelecleucel on Day 1; and IV infusion of tabelecleucel (tab-cel) at 2 x 10^6 T-cells/kg on Days 1, 8, and 15 of each 21-day treatment/consolidation cycles (at least 2 cycles or up to 4 cycles). From the Maintenance Phase, subjects with stable disease or better will receive tabelecleucel on Day 1 and pembrolizumab on Day 1, Day 21, Day 42, and Day 63 of each 84- day maintenance cycle, which was continued until disease progression, unacceptable toxicity, or a total of 35 pembrolizumab infusions (including for treatment, consolidation, and maintenance) had been administered, whichever occurred first.
- Cohort 1B: Checkpoint Inhibitor PD-1/PD-L1 Failure: Checkpoint inhibitor PD-1/PD-L1 failure subjects during the treatment phase received IV infusion of pembrolizumab at 200 mg for adults (≥ 18 years of age) or 2 mg/kg for adolescents (12 to < 18 years of age) prior to the administration of tabelecleucel on Day 1; and IV infusion of tabelecleucel (tab-cel) at 2 x 10^6 T-cells/kg on Days 1, 8, and 15 of each 21-day treatment/consolidation cycles (at least 2 cycles or up to 4 cycles). From the Maintenance Phase, subjects with stable disease or better will receive tabelecleucel on Day 1 and pembrolizumab on Day 1, Day 21, Day 42, and Day 63 of each 84-day maintenance cycle, which was continued until disease progression, unacceptable toxicity, or a total of 35 pembrolizumab infusions (including for treatment, consolidation, and maintenance) had been administered, whichever occurred first.
- Cohort 2: Checkpoint Inhibitor Naïve: Checkpoint inhibitor naive subjects during the treatment phase received IV infusion of pembrolizumab at 200 mg for adults (≥ 18 years of age) or 2 mg/kg for adolescents (12 to < 18 years of age) prior to the administration of tabelecleucel on Day 1; and IV infusion of tabelecleucel (tab-cel) at 2 x 10^6 T-cells/kg on Days 1, 8, and 15 of each 21-day treatment/consolidation cycles (at least 2 cycles or up to 4 cycles). From the Maintenance Phase, subjects with stable disease or better will receive tabelecleucel on Day 1 and pembrolizumab on Day 1, Day 21, Day 42, and Day 63 of each 84- day maintenance cycle, which was continued until disease progression, unacceptable toxicity, or a total of 35 pembrolizumab infusions (including for treatment, consolidation, and maintenance) had been administered, whichever occurred first.
Period: Overall Study
Arm/Group | Cohort 1B: Checkpoint Inhibitor Naïve | Cohort 1B: Checkpoint Inhibitor PD-1/PD-L1 Failure | Cohort 2: Checkpoint Inhibitor Naïve
Started | 6 | 6 | 0
Completed | 0 | 0 | 0
Not Completed | 6 | 6 | 0
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Death | 3 | 3 | 0
Not completed — Study Terminated By Sponsor | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all participants who received at least 1 dose of investigational products (tabelecleucel or pembrolzumab). No participants were enrolled in Phase 2 (Cohort 2) due to early study termination.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1B: Checkpoint Inhibitor Naïve | Cohort 1B: Checkpoint Inhibitor PD-1/PD-L1 Failure | Cohort 2: Checkpoint Inhibitor Naïve | Total
Number analyzed (Participants) | 6 | 6 | 0 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.0 (16.97) | 53.0 (3.16) |  | 51.0 (11.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 0 | 6
  Male | 2 | 4 | 0 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 0 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 5 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 1 | 1 | 0 | 2
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1B: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: The occurrence of any of the following toxicities during Treatment Cycle 1 will be considered a DLT, if assessed by the investigator to be possibly related or related to investigational product administration (either tabelecleucel and/or pembrolizumab): Grade (G) 4 nonhematologic toxicity; G4 hematologic toxicity lasting >=7 days, except thrombocytopenia; any nonhematologic AE >=G3, except G3 fatigue lasting =<3 days; G3 diarrhea, nausea, or vomiting; G3 rash; Any G3/4 non-hematologic laboratory value if clinically significant medical intervention is required to treat the participant, abnormality leads to hospitalization, abnormality persists for > 1 week, abnormality results in a Drug-induced Liver Injury (DILI); G3/4 febrile neutropenia; > 2 weeks delay in initiating Cycle 2; discontinue treatment during Cycle 1; missing > 25% of study drugs doses as a result of investigational product-related AEs during the first cycle;G5 toxicity.
Time Frame: From Day 1 through Day 21 of Cycle 1
Population: Full analysis set included all participants who received at least one dose of investigational products (tabelecleucel or pembrolizumab) and were observed during the first 21 days of the first cycle.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1B: Checkpoint Inhibitor Naïve: Checkpoint inhibitor naive subjects during the treatment phase received IV infusion of pembrolizumab at 200 mg for adults (≥ 18 years of age) or 2 mg/kg for adolescents (12 to < 18 years of age) prior to the administration of tabelecleucel on Day 1; and IV infusion of tabelecleucel (tab-cel) at 2 x 10^6 T-cells/kg on Days 1, 8, and 15 of each 21-day treatment/consolidation cycles (at least 2 cycles or up to 4 cycles). From the Maintenance Phase, subjects with stable disease or better will receive tabelecleucel on Day 1 and pembrolizumab on Day 1, Day 21, Day 42, and Day 63 of each 84- day maintenance cycle, which was continued until disease progression, unacceptable toxicity, or a total of 35 pembrolizumab infusions (including for treatment, consolidation, and maintenance) had been administered, whichever occurred first.
Arm/Group | Cohort 1B: Checkpoint Inhibitor Naïve | Cohort 1B: Checkpoint Inhibitor PD-1/PD-L1 Failure
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

2. Primary Outcome: Cohort 1B: Maximum Tolerated Dose (MTD)
Description: The MTD is defined as the highest dose level at which the subject incidence of a DLTs during the first 21-day cycle of investigational product dosing is < 33%
Time Frame: From Day 1 through Day 21 of Cycle 21
Population: The study was terminated before the outcome measure data were collected, refer to the Limitations and Caveats section for additional information.
Arm/Group | Cohort 1B: Checkpoint Inhibitor Naïve | Cohort 1B: Checkpoint Inhibitor PD-1/PD-L1 Failure
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Cohort 1B: Recommended Phase 2 Dose (RP2D) of Tabelecleucel in Combination With Pembrolizumab
Description: The RP2D is no higher than the maximum tolerated dose (highest dose level at which the number of participants with a DLTs during the first 21-day cycle of investigational product dosing is < 33%) and is based on optimal benefit-risk, as determined by the Safety Data Review Committee (SDRC).
Time Frame: From Day 1 through Day 21 of Cycle 1
Population: as for outcome 1
Measure: Number; unit: cells/kg
Groups:
- Cohort 1B: Checkpoint Inhibitor Naïve and PD-1/PD-L1 Failure: Checkpoint inhibitor naive and PD-1/PD-L1 failure subjects during the treatment phase received IV infusion of pembrolizumab at 200 mg for adults (≥ 18 years of age) or 2 mg/kg for adolescents (12 to < 18 years of age) prior to the administration of tabelecleucel on Day 1; and IV infusion of tabelecleucel (tab-cel) at 2 x 10^6 T-cells/kg on Days 1, 8, and 15 of each 21-day treatment/consolidation cycles (at least 2 cycles or up to 4 cycles). From the Maintenance Phase, subjects with stable disease or better will receive tabelecleucel on Day 1 and pembrolizumab on Day 1, Day 21, Day 42, and Day 63 of each 84- day maintenance cycle, which was continued until disease progression, unacceptable toxicity, or a total of 35 pembrolizumab infusions (including for treatment, consolidation, and maintenance) had been administered, whichever occurred first.
Arm/Group | Cohort 1B: Checkpoint Inhibitor Naïve and PD-1/PD-L1 Failure
Number analyzed (Participants) | 12
cells/kg | 2000000

4. Primary Outcome: Cohort 1B: Characterization of the Safety Profile: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as any AE occurring after initiation of the first dose of study treatment through 30 days after the last administration of study drugs or any pre-existing AE (ie, started prior to the first dose of study drugs) that worsened after the first dose through 30 days after the last administration of study drugs or any related AE on or after first dose.
Time Frame: From Day 1 to end of study (1 year after the last dose or until disease progression, whichever occurred first) (approximately 27 months)
Population: Full analysis set included all participants who received at least one dose of investigational products (tabelecleucel or pembrolizumab).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1B: Checkpoint Inhibitor Naïve | Cohort 1B: Checkpoint Inhibitor PD-1/PD-L1 Failure
Number analyzed (Participants) | 6 | 6
Participants
  Any TEAEs | 6 | 6
  TEAEs (worst grade >=3) | 1 | 4
  TEAEs fatal | 0 | 0
  TEAEs leading to treatment interruption | 0 | 0
  TEAEs leading to treatment discontinuation | 4 | 4
  Any TESAEs | 1 | 1
  TEAEs related or possibly related to study treatment (worst grade >=3) | 0 | 0
  TEAEs related or possibly related to study treatment; serious | 0 | 1
  TEAEs related or possibly related to study treatment; fatal | 0 | 0
  TEAEs related or possibly related to study treatment; leading to treatment interruption | 0 | 0
  TEAEs related or possibly related to study treatment; leading to treatment discontinuation | 0 | 0

5. Primary Outcome: Cohort 2: Characterization of the Safety Profile: Number of Participants With TEAEs and TESAEs
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as any AE occurring after initiation of the first dose of study treatment through 30 days after the last administration of study drugs or any pre-existing AE (ie, started prior to the first dose of study drugs) that worsened after the first dose through 30 days after the last administration of study drugs or any related AE on or after first dose
Time Frame: as for outcome 4
Population: The study did not proceed to Cohort 2 (Phase 2) and data were not collected.
Arm/Group | Cohort 2: Checkpoint Inhibitor Naïve
Number analyzed (Participants) | 0

6. Primary Outcome: Cohort 2: Objective Response Rate (ORR)
Description: For this study, radiographic tumor assessment was performed by computed tomography (CT) or magnetic resonance imaging (MRI) scan based on Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1) and immune RECIST (iRECIST) criteria. Per RECIST v1.1, ORR is defined as percentage of participants with complete response (CR) (disappearance of all extranodal target lesions and all pathological lymph nodes must have decreased to <10 mm in short axis) or partial response (PR) (at least a 30% decrease in sum of the longest diameters of target lesions taking as reference baseline sum diameters). Per iRECIST, immune complete response (iCR) is defined as resolution of all lesions and immune partial response (iPR) is defined as the target lesion sum of diameters (initial target lesions) not above initial progressive disease threshold, no significant growth in non-target lesion overall, and no new lesion or appearance of any new factor.
Time Frame: as for outcome 4
Population: The study did not proceed to Cohort 2 (Phase 2) and data were not collected.
Arm/Group | Cohort 2: Checkpoint Inhibitor Naïve
Number analyzed (Participants) | 0

7. Secondary Outcome: Cohort 2: Complete Response (CR) Rate
Description: The CR rate is defined as percentage of participants with complete response. Per RECIST v1.1, CR is defined as disappearance of all extranodal target lesions and all pathological lymph nodes must have decreased < 10 mm in short axis.
Time Frame: as for outcome 4
Population: The study did not proceed to Cohort 2 (Phase 2) and data were not collected.
Arm/Group | Cohort 2: Checkpoint Inhibitor Naïve
Number analyzed (Participants) | 0

8. Secondary Outcome: Cohort 2: Duration of Response (DOR)
Description: Per RECIST v1.1, the DoR is defined as the time from the date of first documented confirmed response until date of documented progression or death in the absence of disease progression.
Time Frame: as for outcome 4
Population: The study did not proceed to Cohort 2 (Phase 2) and data were not collected.
Arm/Group | Cohort 2: Checkpoint Inhibitor Naïve
Number analyzed (Participants) | 0

9. Secondary Outcome: Cohort 2: Progression Free Survival (PFS)
Description: The PFS is defined as the time from the first dose of investigational product until the date of RECIST v1.1 defined progression or death due to any cause, whichever occurred first.
Time Frame: as for outcome 4
Population: The study did not proceed to Cohort 2 (Phase 2) and data were not collected.
Arm/Group | Cohort 2: Checkpoint Inhibitor Naïve
Number analyzed (Participants) | 0

10. Secondary Outcome: Cohort 2: Overall Survival (OS)
Description: The OS is defined as the time from the first dose of investigational product to the date of death due to any cause.
Time Frame: as for outcome 4
Population: The study did not proceed to Cohort 2 (Phase 2) and data were not collected.
Arm/Group | Cohort 2: Checkpoint Inhibitor Naïve
Number analyzed (Participants) | 0

11. Secondary Outcome: Cohort 2: Immune Response Rate (iRR)
Description: iRR is iCR + iPR. Per iRECIST, iCR is defined as resolution of all lesions and iPR is defined as the target lesion sum of diameters (initial target lesions) not above initial progressive disease threshold, no significant growth in non-target lesion overall, and no new lesion or appearance of any new factor.
Time Frame: as for outcome 4
Population: The study did not proceed to Cohort 2 (Phase 2) and data were not collected.
Arm/Group | Cohort 2: Checkpoint Inhibitor Naïve
Number analyzed (Participants) | 0

12. Secondary Outcome: Cohort 2: Duration of Immune Response (DOiR)
Description: DOiR is duration of iCR + iPR. Per iRECIST, iCR is defined as resolution of all lesions and iPR is defined as the target lesion sum of diameters (initial target lesions) not above initial progressive disease threshold, no significant growth in non-target lesion overall, and no new lesion or appearance of any new factor.
Time Frame: as for outcome 4
Population: The study did not proceed to Cohort 2 (Phase 2) and data were not collected.
Arm/Group | Cohort 2: Checkpoint Inhibitor Naïve
Number analyzed (Participants) | 0

13. Post Hoc Outcome: Cohort 1B: Objective Response Rate (ORR)
Description: For this study, radiographic tumor assessment was performed by CT or MRI scan based on RECIST v1.1 and iRECIST criteria. Per RECIST v1.1, ORR is defined as percentage of participants with CR (disappearance of all extranodal target lesions and all pathological lymph nodes must have decreased to <10 mm in short axis) or PR (at least a 30% decrease in sum of the longest diameters of target lesions taking as reference baseline sum diameters). Per iRECIST, iCR is defined as resolution of all lesions and iPR is defined as the target lesion sum of diameters (initial target lesions) not above initial progressive disease threshold, no significant growth in non-target lesion overall, and no new lesion or appearance of any new factor. Refer also to the Limitations and Caveats section.
Time Frame: as for outcome 4
Population: Full analysis set included all participants who received at least one dose of investigational products (tabelecleucel or pembrolizumab). Cohort 1B (Phase 1b) was not powered for efficacy.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1B: Checkpoint Inhibitor Naïve | Cohort 1B: Checkpoint Inhibitor PD-1/PD-L1 Failure
Number analyzed (Participants) | 6 | 6
Percentage of Participants | 0 [0.0 to 45.9] | 0 [0.0 to 45.9]

14. Post Hoc Outcome: Cohort 1B: Clinical Benefit Rate (CBR)
Description: The CBR is defined as the proportion of subjects who achieved BOR of CR or PR or SD. CR and PR are defined in outcome measure of ORR. The SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. For this study, radiographic tumor assessment was performed by CT scan or MRI scan based on RECIST v1.1 and immune-based RECIST criteria. Refer also to the Limitations and Caveats section.
Time Frame: as for outcome 4
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort 1B: Checkpoint Inhibitor Naïve | Cohort 1B: Checkpoint Inhibitor PD-1/PD-L1 Failure
Number analyzed (Participants) | 6 | 6
Percentage of Participants | 66.7 [22.3 to 95.7] | 33.3 [4.3 to 77.7]

ADVERSE EVENTS:
Time Frame: From Day 1 to end of study (1 year after the last dose or until disease progression, whichever occurred first) (approximately 27 months)
Description: No participants were enrolled in phase 2 (cohort 2) due to early study termination, so, number of participants at risk for All-cause mortality, serious adverse events, and other (not including serious) adverse events are zero.
Arm/Group | Cohort 1B: Checkpoint Inhibitor Naïve | Cohort 1B: Checkpoint Inhibitor PD-1/PD-L1 Failure | Cohort 2: Checkpoint Inhibitor Naïve
All-Cause Mortality (participants affected / at risk) | 3/6 | 3/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/6 | 0/0
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1B: Checkpoint Inhibitor Naïve (N=6) | Cohort 1B: Checkpoint Inhibitor PD-1/PD-L1 Failure (N=6) | Cohort 2: Checkpoint Inhibitor Naïve (N=0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1B: Checkpoint Inhibitor Naïve (N=6) | Cohort 1B: Checkpoint Inhibitor PD-1/PD-L1 Failure (N=6) | Cohort 2: Checkpoint Inhibitor Naïve (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (3) | 1 (1) | 0 (0)
Blindness unilateral (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (4) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 1 (2) | 0 (0)
Chills (General disorders) | 2 (3) | 0 (0) | 0 (0)
Disease progression (General disorders) | 5 (5) | 3 (3) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (5) | 0 (0)
Fatigue (General disorders) | 2 (4) | 1 (3) | 0 (0)
Nodule (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 2 (7) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (2) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (2) | 0 (0)
Serum ferritin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (5) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Facial motor skill dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin tightness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Post-Hoc efficacy outcomes (ORR and CBR) were analyzed for Cohort 1B (phase 1); however, Cohort 1B was not powered for efficacy. The study was deprioritized and terminated early, and did not proceed to Cohort 2 (Phase 2).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/67/NCT03769467/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/67/NCT03769467/SAP_001.pdf